CLINICAL TRIAL: NCT01578005
Title: Intravascular Ultrasound (IVUS) Assessment of the Atherosclerotic Plaque Causing an Acute Coronary Syndrome: One-year Changes Under Optimal Secondary Prevention Drug Treatment
Brief Title: IVUS Assessment of Atheroma Burden After Acute Coronary Syndrome
Acronym: OPTIVUS
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/10/047; 2010-A00471-38 (Other: ANSM)
Record Dates: First submitted 2011-06-30; First posted 2012-04-16 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; IVUS; atherosclerotic plaque
MeSH Terms: conditions — Acute Coronary Syndrome; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bioanalysis on DNA, searching genes involving coronary disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary angioplasty is rather frequently performed in such situations, presumably because, changes in the atherosclerotic plaque under drug treatment, have remained poorly described so far. Intravascular ultrasound (IVUS) enables a precise description of coronary atheroma, better than the one provided by coronary angiography.

DETAILED DESCRIPTION:
According to current guidelines, patients with coronary lesions with stenosis <70% should receive optimal secondary prevention drug treatment without angioplasty, even after an acute coronary syndrome (ACS). Nevertheless, coronary angioplasty is rather frequently performed in such situations, presumably because, changes in the atherosclerotic plaque under drug treatment, have remained poorly described so far. Intravascular ultrasound (IVUS) enables a precise description of coronary atheroma, better than the one provided by coronary angiography.

The first objective is to assess by endo-coronary ultrasound, under optimal medical treatment, the evolution of atheromatous plaque (with stenosis <70%). The evolution will be appreciated after 12 months of treatment the percentage of atheromatous volume (PVA). The aim of the first secondary objective to evaluate, after 12 months of treatment, the evolution of the total atheromatous volume (VAT) and the standardized total atheromatous volume (standardized VAT). The Second secondary objective is to evaluate by endo-coronary ultrasound, the evolution of a stable atheromatous plaque. This analysis will be performed in patients with a second coronary lesion (atheroma plaque), resulting in less than 70% stenosis, and not being responsible for acute coronary syndrome. The evolution of the stable plate will be compared to the evolution of the unstable plate. Finally, the third secondary objective is to estimate the incidence of clinical events (death, acute coronary syndromes, ischemic stroke, revascularization, hospitalization for heart failure) within 12 months of the occurrence of an acute coronary syndrome managed by medical treatment optimal secondary prevention (without performing angioplasty).

ELIGIBILITY:
Inclusion Criteria:

* adult patients hospitalized for ACS, for whom the target lesion has less than 70% stenosis and not treated with coronary angioplasty.

Exclusion Criteria:

* Patients presenting with a target lesion with ≥70% stenosis ; Patients for whom the target lesion is treated with coronary angioplasty ; Interventions: A first IVUS will be performed after the acute coronary event (baseline) and will be done again one-year after to assess changes in the atherosclerotic plaques.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female and male aged more than 18 years hospitalized for acute coronary syndrom
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
atheroma volume | one year
  One-year changes in percent atheroma volume (PAV), measured in the lesion which has promoted the ACS (unstable plaque).

SECONDARY OUTCOMES:
PAV | 1 year
  One-year changes total atheroma volume (TAV) and normalized TAV. One year changes in PAV, TAV and normalized TAV in a stable plaque (not involved in the ACS).
incidence of the clinical cardiovascular events | 1 year
  one year incidence of clinical cardiovascular events (death, acute coronary syndrome, ischaemic stroke, revascularization, hospitalization for heart failure).
TAV | 1 year
  One-year changes in PAV, TAV and normalized TAV, in a stable plaque (not involved in the ACS)
normalized TAV | 1 year
  One-year changes in PAV, TAV and normalized TAV, in a stable plaque (not involved in the ACS)

CONTACTS AND LOCATIONS:
Overall Officials: Meyer Elbaz, PhD, Study Chair — University Hospital, Toulouse; Pierre Coste, PhD, Principal Investigator — University Hospital, Bordeaux; Patrice Virot, PhD, Principal Investigator — UH Limoges
Locations (3):
- France (3):
  - UH Bordeaux Haut-Lévêque, Pessac, Bordeaux Pessac
  - UH Limoges, Limoges
  - UH Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No